CLINICAL TRIAL: NCT07099209
Title: The Use of Delta-Wave Hypnosis as a Non-Pharmacological Adjunct to Reduce Perioperative Anxiety During Cataract Surgery: A Prospective, Randomized, Single-Blind Study
Brief Title: Delta-Wave Hypnoanalgesia for Reducing Perioperative Anxiety in Cataract Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Military Hospital of Tunis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Military-Hypno-CAT-2023
Record Dates: First submitted 2025-07-18; First posted 2025-08-01 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-08

CONDITIONS: Cataract; Anxiety
Keywords: Cataract Surgery; Perioperative Anxiety; Hypnosis; Audioanalgesia; Delta-Wave Stimulation
MeSH Terms: conditions — Cataract; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypnosis Group (Experimental): Patients received delta-wave binaural beats via headphones starting 15 minutes before surgery and continuing intraoperatively.
  Interventions: Behavioral: Delta-Wave Hypnoanalgesia
- Control Group (No Intervention): Patients received standard care with no auditory intervention.

INTERVENTIONS:
Behavioral: Delta-Wave Hypnoanalgesia — Binaural beat audio tracks at delta frequencies (1-4 Hz) to induce deep relaxation and reduce perioperative anxiety.
  Arms: Hypnosis Group

SUMMARY:
This prospective, randomized, single-blind trial evaluated the effect of delta-wave binaural beat audio hypnoanalgesia, a non-pharmacological hypnosis technique, on reducing perioperative anxiety and improving hemodynamic stability during cataract surgery performed under local anesthesia. A total of 198 patients were randomized into two groups: one group received delta-wave auditory stimulation, while the control group received standard care without auditory intervention. The primary outcomes measured included changes in anxiety levels, assessed using the Amsterdam Preoperative Anxiety and Information Scale (APAIS), as well as heart rate and blood pressure parameters.

DETAILED DESCRIPTION:
This prospective interventional study aimed to assess the efficacy of delta-wave auditory hypnoanalgesia, a non-pharmacological adjunct technique, during cataract surgery performed under regional anesthesia. Patients in the hypnosis group received binaural beats with delta-frequency waves through headphones before and during the operation. The control group received no auditory stimulation. Hemodynamic parameters including heart rate (HR), systolic blood pressure (SBP), diastolic blood pressure (DBP), and mean arterial pressure (MAP) were recorded, alongside assessments of anxiety using the Amsterdam Preoperative Anxiety and Information Scale (APAIS), pain measured by the Numeric Rating Scale (NRS), bispectral index (BIS) monitoring, and patient satisfaction scores at various time points. The findings support the anxiolytic effect of delta-wave hypnoanalgesia and suggest its potential role in improving patient comfort and satisfaction during cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75
* Undergoing cataract surgery under locoregional anesthesia
* Provided written informed consent

Exclusion Criteria:

* Hearing impairment
* Cognitive disorders
* Requirement for general anesthesia or sedation
* Refusal to participate

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2023-09-28 (Actual); Primary Completion 2024-01-12 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
Amsterdam Preoperative Anxiety and Information Scale (APAIS) | Baseline to start of surgery
  The total anxiety score ranges from 4 to 20. Higher scores indicate higher levels of preoperative anxiety.

SECONDARY OUTCOMES:
Intraoperative heart rate variation | Every 5 minutes throughout the surgical procedure
  Heart rate will be recorded at 5-minute intervals during the surgery. Variations in heart rate will be analyzed as an indicator of autonomic response to anxiety and hypnoanalgesia. Lower or more stable values may reflect a calming effect.
Intraoperative blood pressure changes | Intraoperative period (every 5 minutes throughout the surgery)
  Systolic, diastolic, and mean arterial pressure (SBP, DBP, MAP) measured every 5 minutes during surgery.
Numeric Rating Scale (NRS) for pain | Throughout the surgical procedure (intraoperative period)
  Ranging from 0 to 10. A score of 0 indicates "no pain," while a score of 10 indicates "the worst pain imaginable." Higher scores indicate worse pain perception.
Bispectral Index Score (BIS) | Throughout the surgical procedure
  ranging from 0 to 100. Values below 60 indicate deep sedation, while values between 61 and 90 indicate moderate sedation to mild anxiolysis. Higher scores indicate higher levels of consciousness (less sedation).
Satisfaction score from patient, surgeon, and anesthesiologist (0-10 scale) | Immediately after surgery (Day 0)
  Numerical scale from 0 (minimum) to 10 (maximum). Higher scores reflect greater satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Main Military Hospital of Tunis, Tunis, Montfleury, Tunisia

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to concerns related to patient privacy and confidentiality, as well as restrictions imposed by ethical approvals and informed consent agreements. Additionally, there may be legal and institutional policies limiting data sharing. We are committed to protecting participant identities and complying with all regulatory requirements.

DOCUMENTS (3):
  • Study Protocol (2023-09-15): https://cdn.clinicaltrials.gov/large-docs/09/NCT07099209/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-15): https://cdn.clinicaltrials.gov/large-docs/09/NCT07099209/SAP_001.pdf
  • Informed Consent Form (2023-09-15): https://cdn.clinicaltrials.gov/large-docs/09/NCT07099209/ICF_002.pdf